CLINICAL TRIAL: NCT01463215
Title: An Open-Label, Dose Escalation With 2 Dose Levels, Proof-of-Concept Clinical Trial of Ambroxol for the Treatment of Type I Gaucher Disease
Brief Title: Clinical Trial of Ambroxol in Patients With Type I Gaucher Disease
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Exsar Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-Ambroxol-002
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Type I Gaucher Disease
Keywords: Ambroxol; Type I Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Ambroxol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ambroxol (Experimental): Ambroxol at a dose level of 187.5 or 225 mg/day will be given once daily by mouth for 2 months.
  Interventions: Drug: Ambroxol

INTERVENTIONS:
Drug: Ambroxol — Ambroxol at a dose level of 187.5 or 225 mg/day will be given once daily by mouth for 2 months.
  Other Names: Mucosolvon®

SUMMARY:
Ambroxol is expected to improve the signs and symptoms of patients with Type I Gaucher Disease.

DETAILED DESCRIPTION:
This is an Open-Label, Dose Escalation with 2 Dose Levels, Proof-of-Concept Clinical Trial of Ambroxol for the Treatment of Patients with Type I Gaucher Disease.

This study is a randomized clinical trial involving 20 evaluable patients affected with Type 1 Gaucher disease who are responsive to Ambroxol in vitro. There are 2 treatment groups, involving 2 dose levels of Ambroxol (187.5 and 225 mg/day), given once daily PO for 2 months in both groups. The 187.5-mg/day dose level will be tested first. If there are no significant adverse events, defined as >Grade 3 toxicity according to the latest version of the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), the 225-mg/day dose level will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and genetically confirmed diagnosis of Gaucher disease caused by β-glucocerebrosidase deficiency resulting from mutations in the GBA genes, which have been shown to respond to Ambroxol according to in vitro screening assay.
* Must be 16 years of age or older at the time of study initiation.
* With an intact, enlarged spleen.
* A hemoglobin level of at least 10 g/L.
* Able to understand and cooperate with the requirements of the study protocol.
* Mentally competent, have ability to understand and willingness to sign the informed consent form.
* Able to travel to a participating study site.
* Women of child-bearing potential must use accepted contraceptive methods, and must have a negative serum or urine pregnancy test within one week prior to treatment initiation. An additional pregnancy test is to be performed, and results obtained, prior to administration of the first dose of Ambroxol.
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists.
* Body weight >40 kg (88 lbs).

Exclusion Criteria:

* Receipt of any form of glucocerebrosidase <<4 weeks prior study initiation.
* Total splenectomy.
* Serious medical illness, significant cardiac disease, chronic bronchitis, emphysema, and cystic fibrosis, as well as disorders causing ventilation perfusion mismatch.
* Substance abuse.
* Any complex disease that may confound treatment assessment.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception.
* Lactating females because of the potential for adverse reactions in nursing infants.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Unwilling or unable to follow protocol requirements.
* Known hypersensitivity reactions, intolerance or adverse reactions to Ambroxol or to the inactive ingredients.
* Evidence of systemic infection, or serious infection within the past month.
* Known to have HIV infection.
* Known to have hepatitis B or hepatitis C.
* Patients with a history of convulsive disorders.
* Patients receiving any other investigational treatment for any indication within the past 4 weeks prior to initiation of Ambroxol treatment.
* A history of cancer of any type.
* Patients who have received immunotherapy of any type within the past 4 weeks prior to study initiation.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Safety assessment based on potential changes in physical exam, vital signs, ECG, adverse event query, and clinical lab results, when compared to baseline values. | Safety will be assessed at baseline and biweekly for 2 months.
  Safety will be based on physical exam, vital signs, ECG, adverse event query, and clinical pathology (includes chemistry, hematology and coagulation), asessed at baseline and approximately biweekly during the study.

SECONDARY OUTCOMES:
efficacy based on biomarker (glucocerebrosidase activities), lab results, as well as hepatic and splenic volumes from imaging scans. | Biomarker, lab results (phenotype), as well as hepatic and spenic volumes will be assessed at baseline and after 2 months of treatment, and lab results (phenotypes) will also be assessed biweekly during the 2-month treatment period.
  Efficacy is based on biomarker (glucocerebrosidase activities), phenotypes according to specific lab results (acid phosphatase, angiotensin-converting enzyme, serum bilirubin, hemoglobin, platelet counts, peripheral blood leukocyte counts, serum iron, clotting time, etc.), as well as hepatic and splenic volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Johnston, Study Chair — Exsar Corporation
Locations (1):
- ExSAR Corporation, Monmouth Junction, New Jersey, United States